CLINICAL TRIAL: NCT06911671
Title: Innovative Upper Limb Stroke Rehabilitation Approach Combining Myoelectric Control Assistance in Virtual Reality and Cerebellar TBS Plasticity Enhancement
Brief Title: EMG Control Assistance Virtual Reality Interface Coupled With Cerebellar-iTBS for Arm Recovery After Stroke (ERICA)
Acronym: ERICA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: I.R.C.C.S. Fondazione Santa Lucia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PROG.899; GR-2019-12370271 (Other Grant/Funding Number: Italian Ministry of Health)
Record Dates: First submitted 2023-02-03; First posted 2025-04-04 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2025-03

CONDITIONS: Stroke; Stroke, Cardiovascular
Keywords: Virtual Reality; Brain Stimulation; Myoelectric Control; Transcranial Magnetic Stimulation; Cerebellar Stimulation; Motor Recovery; Tailored Assistance
MeSH Terms: conditions — Stroke; Myocardial Infarction | interventions — Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- EMG-VR real c-iTBS (Experimental): Subjects will perform 12 sessions (~30 minutes, 3 times per weeks for 4 weeks) of assisted EMG control task (aEC) after real cerebellar intermittent theta burst stimulation (c-iTBS) for paretic upper limb.
  Interventions: Device: Virtual Reality Interface + Cerebellar iTBS (c-iTBS)
- EMG-VR sham c-iTBS (Sham Comparator): Subjects will perform 12 sessions (~30 minute, 3 times per weeks for 4 weeks) of assisted EMG control task (aEC) after sham cerebellar intermittent theta burst stimulation (c-iTBS) for paretic upper limb.
  Interventions: Device: Virtual Reality + Sham Cerebellar iTBS (sham c-iTBS)
- Conventional Physical Therapy (Active Comparator): Subjects will perform 12 sessions (~30 minutes, 3 times per weeks for 4 weeks) of physical therapy targeting on motor functionality of upper limb.
  Interventions: Other: Physical Therapy

INTERVENTIONS:
Device: Virtual Reality Interface + Cerebellar iTBS (c-iTBS) — Subjects will sit in a chair with their forearm inserted in a splint attached to a force transducer. The subjects' view of their hand will be occluded by a mirror displaying the virtual scene. EMGs from arm and shoulder muscles will be recorded by surface EMG electrodes. Subjects will displace a virtual handle according to either the forces recorded by the force transducer or forces estimated from the recorded EMGs (EMG control).
  Arms: EMG-VR real c-iTBS
Device: Virtual Reality + Sham Cerebellar iTBS (sham c-iTBS) — c-iTBS will be carried out using Magstim Rapid magnetic biphasic stimulator. Twenty 2-s trains of three-pulse bursts at 50 Hz repeated every 200 ms with an inter-train interval of 10 s, for a total of 190 s will be applied over the contralesional lateral cerebellum. The coil will be positioned tangentially to the scalp for real and 90° angled for sham c-iTBS.
  Arms: EMG-VR sham c-iTBS
Other: Physical Therapy — Passive mobilization and motor recruitment of impaired upper limb will be performed with the support of a physical therapist specialized in neurological rehabilitation.
  Arms: Conventional Physical Therapy

SUMMARY:
The investigators hypothesize that a myoelectric (EMG) controlled virtual reality (VR) interface allows for effective upper limb motor recovery of stroke patients. EMG control offers the possibility to alter visual feedback according to the recorded muscle activity in real-time. By manipulating the motion of a virtual hand associated with the recorded muscle patterns, assistance can be provided to stroke patients by correcting the error between the actual (dysfunctional) and a reference (functional) muscle pattern. Thus, through such an assistive EMG control algorithm, patients will be able to perform reaching movements with the virtual hand despite their motor impairment. By gradually reducing assistance, it is hypothesized that the salient error in the task space provided as visual feedback will systematically change the muscle patterns, thereby driving adaptation of the dysfunctional muscle patterns, enhancing motor recovery. Moreover, due to its relevant role in motor learning, it is expected that cerebellar stimulation will favor the underlying processes of adapting cerebello-cortical plasticity involved in motor learning. Therefore, it is hypothesized that an assistive EMG control algorithm in combination with cerebellar transcranial magnetic stimulation will further enhance upper limb recovery.

DETAILED DESCRIPTION:
Theta burst stimulation (TBS) is a novel form of repetitive transcranial magnetic stimulation that mimics protocols inducing long-term potentiation (LTP) or long-term depression. Theta burst stimulation (TBS) is a novel form of repetitive transcranial magnetic stimulation that mimics protocols inducing long-term potentiation (LTP) or long-term depression (LTD) in animal models. Whereas continuous TBS induces long-lasting inhibition of cortical areas, iTBS exerts the opposite effect, increasing cerebellar excitability.

ELIGIBILITY:
Inclusion Criteria:

* First ever ischemic stroke with mild to moderate motor impairment of upper limb;
* Left or right sub-cortical or cortical lesion of the middle cerebral artery;
* Age>18, <80 years;
* No visuospatial, cognitive, or attention deficits;
* Fugl-Meyer score<56.

Exclusion Criteria:

* History of seizures;
* Treatment with Benzodiazepines, Baclofen;
* Pregnancy status;
* Intracranial metal implant;
* Cardiac pace-maker;
* Orthopedic upper limb limitation;
* Upper limb pain;
* Patients with neurological diseases beyond stroke or with neuropsychiatric disorders or with neuropsychological disorders that could potentially compromise informed consent or compliance during the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2027-08-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
Change in the Fugl-Meyer Assessment Scale for Upper Extremity (FMA-UE) | baseline: T0, post-treatment (3 weeks): T1, follow-up (6 weeks from T1): T2.
  Comprehensive clinical measurement tool of upper limb functions after stroke. Range score form 0 to 66 points, a higher score represents an improvement.

SECONDARY OUTCOMES:
Change in the Box and Block test (BBT) | baseline: T0, post-treatment (3 weeks): T1, follow-up (6 weeks from T1): T2.
  BBT assesses the patient's manual dexterity. It is composed of a wooden box divided into two compartments by a partition and 150 blocks. The BBT administration consists of asking the client to move, one by one, the maximum number of blocks from one compartment of the box to the other of equal size within 60 seconds. The test is performed with both upper limbs separately to evaluate the manual dexterity of each arm individually.
Change in modified Barthel Index (mBI) score | baseline: T0, post-treatment (3 weeks): T1, follow-up (6 weeks from T1): T2.
  mBI is an ordinal scale that measures functional independence in the domains of personal care and mobility. Score range is from 0 (totally dependent) to 100 (independent).
Change in the Nine Hole Peg Test (NHPT) | baseline: T0, post-treatment (3 weeks): T1, follow-up (6 weeks from T1): T2.
  NHPT assesses the patient's fine manual dexterity and hand-eye coordination. It consists of a small board with nine holes and nine pegs. During the test, the patient is asked to place the pegs into the holes one by one and then remove them as quickly as possible. The total time to complete the task is recorded. The test is performed separately with each upper limb to evaluate the dexterity of both hands individually.
Change in muscle activation patterns (EMG) | baseline: T0, post-treatment (3 weeks): T1, follow-up (6 weeks from T1): T2.
  Task performance in the EMG-control mode will be quantified by the initial angle error and the fraction of unsuccessful trials during the task execution. To combine the initial angle error and the fraction of unsuccessful trials into a single performance index, a linear combination approach will be used. We will compare the initial, baseline performance measure of EMG index of the first session with the performance of the last session.
Change in force-control | baseline: T0, post-treatment (3 weeks): T1, follow-up (6 weeks from T1): T2.
  The change in force-control will be measured using EMG by analyzing the amplitude of the electromyographic signal (EMG) during the task. An increase in EMG amplitude indicates greater muscle activation, which correlates with improved muscle strength. We will compare the initial, baseline measure of force control of the first session with the measure of the last session.
Change in Motor Evoked Potentials' (MEP) Amplitude | baseline: T0, post-treatment (3 weeks): T1, follow-up (6 weeks from T1): T2.
  A single pulse transcranial magnetic stimulation will be applied to the primary motor cortex to produce a recordable motor-evoked potentials in contralateral muscles. The peak-to-peak amplitude of MEPs will be used to represent the cortico-spinal excitability. Both hemispheres will be investigated.

CONTACTS AND LOCATIONS:
Overall Officials: Giacomo Koch, Prof., Study Chair — IRCCS Santa Lucia Foundation
Locations (1):
- IRCCS Santa Lucia Foundation, Roma, Rome, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Huang YZ, Edwards MJ, Rounis E, Bhatia KP, Rothwell JC. Theta burst stimulation of the human motor cortex. Neuron. 2005 Jan 20;45(2):201-6. doi: 10.1016/j.neuron.2004.12.033. PMID 15664172
- [Background] Hummel FC, Cohen LG. Non-invasive brain stimulation: a new strategy to improve neurorehabilitation after stroke? Lancet Neurol. 2006 Aug;5(8):708-12. doi: 10.1016/S1474-4422(06)70525-7. PMID 16857577
- [Background] Spampinato D, Celnik P. Deconstructing skill learning and its physiological mechanisms. Cortex. 2018 Jul;104:90-102. doi: 10.1016/j.cortex.2018.03.017. Epub 2018 Mar 27. PMID 29775838
- [Background] Celnik P. Understanding and modulating motor learning with cerebellar stimulation. Cerebellum. 2015 Apr;14(2):171-4. doi: 10.1007/s12311-014-0607-y. PMID 25283180
- [Background] Berger DJ, Gentner R, Edmunds T, Pai DK, d'Avella A. Differences in adaptation rates after virtual surgeries provide direct evidence for modularity. J Neurosci. 2013 Jul 24;33(30):12384-94. doi: 10.1523/JNEUROSCI.0122-13.2013. PMID 23884944
- [Background] Koch G, Bonni S, Casula EP, Iosa M, Paolucci S, Pellicciari MC, Cinnera AM, Ponzo V, Maiella M, Picazio S, Sallustio F, Caltagirone C. Effect of Cerebellar Stimulation on Gait and Balance Recovery in Patients With Hemiparetic Stroke: A Randomized Clinical Trial. JAMA Neurol. 2019 Feb 1;76(2):170-178. doi: 10.1001/jamaneurol.2018.3639. PMID 30476999